CLINICAL TRIAL: NCT03367078
Title: Observational Study on the Use of Transcranial Direct Stimulation in Patients With Disorder of Consciousness, Due to Severe Acquired Brain Injury, to Stimulate Recovery of Consciousness
Brief Title: tDCS in Patients With Disorder of Consciousness Due to Severe Acquired Brain Injury
Status: Terminated | Type: Observational
Why Stopped: Organizational problems, change of research priorities
Sponsor: Montecatone Rehabilitation Institute S.p.A. (Other)
Responsible Party: Sponsor
Other Study IDs: CE-17101
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Consciousness Disorders; Brain Injuries; Vegetative State; Minimally Conscious State; Cognitive Impairment
Keywords: tDCS; transcranial direct current stimulation; acquired brain injury; coma; vigilance
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries; Persistent Vegetative State; Cognitive Dysfunction; Coma | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tDCS cohort: DOC patients treated according to usual care, plus anodal tDCS (prospective cohort)
  Interventions: Device: Anodal tDCS; Other: Usual care
- Historical control cohort: DOC patients treated according to usual care only (retrospective cohort of patients matched for demographic and clinical characteristics, admitted at the Montecatone Rehabilitation Institute no more than 3 years before the introduction of tDCS)
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Anodal tDCS — Anodal tDCS, on L-DLPFC area, is started 2 weeks after admission to the sABI Operative Unit with: one session per day (in the morning), possibly for 5 consecutive days per week (from Monday to Friday), for 2 consecutive weeks. Each tDCS session lasts 20 minutes. Current intensity is 1 mA during the first week, 2 mA in the second week
  Groups: tDCS cohort
Other: Usual care — Usual care of DOC patients

SUMMARY:
The present observational study is aimed at reporting the short-, mid- and long-term outcomes of patients with Disorder of Consciousness (DOC), in Vegetative State (VS) or Minimally Conscious State (MCS), due to a severe Acquired Brain Injury (sABI), after repeated treatments with anodal Transcranial Direct Current Stimulation (tDCS) on Left Dorsolateral Prefrontal Cortex (L-DLPFC), to stimulate recovery of consciousness. The results obtained will also be compared with those of a historical control cohort, before the introduction of tDCS, matched for demographic and clinical characteristics.

DETAILED DESCRIPTION:
Patients surviving sABI resulting in a coma state, thanks to improvements in early intervention and intensive care technologies, in some cases begin to regain vigilance and consciousness within few weeks from the event. In other cases, however, while regaining vigilance, they may continue to present a DOC state. DOC patients, by definition, are unable to communicate and have severe motor, sensory and cognitive deficits. They can be in a Vegetative State (VS), characterized by wakefulness without consciousness, which can favorably evolve in a Minimally Conscious State (MCS).

Although there are currently no evidence-based guidelines on the treatment of DOC patients to facilitate their recovery of consciousness, several studies published in recent years have focused on various pharmacological and non-pharmacological interventions. Among these, there is a non-invasive stimulation technique, the Transcranial Direct Current Stimulation (tDCS), which has long been known for other indications. tDCS affects the neuronal membrane rest potential and is able to neuromodulate cortical excitability. Protocols in the literature describing the use of tDCS in DOC patients envisage anodal stimulation (active electrode) on the L-DLPFC area, with the reference electrode placed on a homologous controlateral area or on the controlateral shoulder. tDCS variants have also been described, both by type of current delivered and by active electrode's positioning, but they are still experimental.

The Montecatone Rehabilitation Institute (a 3rd level Italian hospital, specialized in intensive rehabilitation of sABI and spinal cord injured patients) has recently started adopting tDCS in clinical practice to stimulate recovery of consciousness of VS or MCS, post-sABI, patients. Since it was already known that a single tDCS applications is not sufficient to elicit detectable and durable responses, the Montecatone Institute's protocol envisages anode application on L-DLPFC area in a 20 minute daily session, possibly for 2 consecutive weeks (5 consecutive days per week). For a gradual and safe approach, 1 milliampere (mA) current intensity is applied during the first week, 2 mA during the second week.

The post-sABI DOC patients treated with tDCS at the Montecatone Institute, compared with the known literature, are more homogeneous with regard to the distance of time from the lesional event, moreover tDCS is administered at an earlier stage. The present observational, longitudinal study is aimed therefore at reporting the outcomes of such DOC patients treated with tDCS by evaluating them with functional and cognitive impairment scales, at short-term (at the conclusion of the first and second week of tDCS treatment), medium-term (3 months after the end of the treatment) and long-term (6 months after the end of the treatment). Electroencephalographic (EEG) pattern data will also be collected. The outcome data obtained will be compared with those of a historical control cohort too, matched for demographic and clinical characteristics. The present study aims at covering the lack in the literature of long-term follow-up data too.

It is expected that the results of the present study may be useful to provide concrete indications for planning further research studies aimed at evaluating the effectiveness of different techniques and/or protocols for application of tDCS in post-sABI DOC patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with Disorder of Consciousness, VS (= LCF 2) or MCS (= LCF 3), due to sABI;
* any etiology, with the exception of extensive haemorrhagic lesions;
* stable clinical conditions.

Exclusion Criteria:

* presence of implanted devices (e.g. pacemakers, intrathecal infusers);
* presence of metallic brain implants (clips) or intracranial implants;
* presence of extensive craniotomy involving the area of application of tDCS;
* history of epileptic seizure;
* mechanical ventilation in place;
* history of psychotic disorders;
* severe neurodegenerative pathology;
* pharmacotherapy with Na+ or Ca++ channel blockers (e.g. Carbamazepine) or with N-Methyl-D-aspartate (NMDA) receptor antagonists (e.g. Dextromethorphan);
* pregnancy in progress.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive DOC patients admitted to the sABI Operative Unit of the Montecatone Rehabilitation Institute
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in coma recovery in the tDCS cohort (short- and mid-term outcomes) | Baseline (initial visit); tDCS session 5 (1 week); tDCS closing session 10 (2 weeks); follow-up 1 (1 week after tDCS closing session 10); follow-up 2 (3 months after tDCS closing session 10)
  Assessment by Coma Recovery Scale-Revised (CRS-R) (on-line, where tDCS is administered)
Change in cognitive functioning level in the tDCS cohort (short- and mid-term outcomes) | Baseline (initial visit); tDCS session 5 (1 week); tDCS closing session 10 (2 weeks); follow-up 1 (1 week after tDCS closing session 10); follow-up 2 (3 months after tDCS closing session 10)
  Assessment by Levels of Cognitive Functioning Scale (LCF) (off-line, i.e. where tDCS is administered, immediately after tDCS session)

SECONDARY OUTCOMES:
Change in coma recovery in the tDCS cohort (long-term outcome) | Baseline (initial visit); follow-up 3 (6 months after tDCS closing session 10)
  Assessment by CRS-R scale
Change in cognitive functioning level in the tDCS cohort (long-term outcome) | Baseline (initial visit); follow-up 3 (6 months after tDCS closing session 10)
  Assessment by LCF scale
Change in disability level in the tDCS cohort (short-, mid- and long-term follow-up) | Baseline (initial visit); follow-up 1 (1 week after tDCS closing session 10); follow-up 2 (3 months after tDCS closing session 10); follow-up 3 (6 months after closing session 10)
  Assessment by Rappaport's Disability Rating Scale (DRS)
Change in electroencephalography pattern in the tDCS cohort | Baseline (initial visit); tDCS tDCS closing session 10 (2 weeks)
  Assessment by electroencephalography (EEG) (off-line, i.e. where tDCS is administered, immediately after tDCS session)
Change in coma recovery between the tDCS cohort and the Historical control cohort | Baseline (initial visit); 3 months; 6 months
  Assessment by CRS-R scale
Change in cognitive functioning level between the tDCS cohort and the Historical control cohort | Baseline (initial visit); 3 months; 6 months
  Assessment by LCF scale
Change in disability level between the tDCS cohort and the Historical control cohort | Baseline (initial visit); 3 months; 6 months
  Assessment by DRS scale

CONTACTS AND LOCATIONS:
Overall Officials: Angela Morreale, MD, Principal Investigator — Montecatone Rehabilitation Institute S.p.A.
Locations (1):
- Montecatone Rehabilitation Institute S.p.A., Imola, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided